CLINICAL TRIAL: NCT03002753
Title: Zum Umgang Mit Aufdringlichen Gedanken Bei Der Zwangsstörung - Zwei Behandlungsstrategien im Vergleich
Brief Title: Dealing With Intrusive Thoughts in OCD - a Comparison of Detached Mindfulness and Cognitive Restructuring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christoph-Dornier-Stiftung für Klinische Psychologie (Other)
Collaborators: Universität Münster (Other)
Responsible Party: Principal Investigator, Prof. Dr. Ulrike Buhlmann, Prof. Dr., Universität Münster
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CDS-MS-JR-2016
Record Dates: First submitted 2016-12-14; First posted 2016-12-26 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: OCD; obsessive-compulsive disorder; cognitive therapy; metacognitive therapy; cognitive restructuring; detached mindfulness; comparison; Germany; Muenster; Christoph-Dornier-Stiftung; metacognition
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Cognitive Restructuring

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (3):
- DM (Experimental): Group of patients receiving detached mindfulness (for details, see detailed description of the study)
  Interventions: Behavioral: detached mindfulness
- CR (Active Comparator): Group of patients receiving cognitive restructuring (for details, see detailed description of the study)
  Interventions: Behavioral: cognitive restructuring
- WL (No Intervention): Waitlist control group, which, however, is again randomized after the waiting time in order to receive one of the two interventions (DM or CR).

INTERVENTIONS:
Behavioral: detached mindfulness — Please see detailed study description.
  Arms: DM
Behavioral: cognitive restructuring — Please see detailed study description.
  Arms: CR

SUMMARY:
The purpose of this study is to assess and compare the overall efficacy and differential effects of detached mindfulness and cognitive restructuring in the treatment of patients with obsessive-compulsive disorder.

DETAILED DESCRIPTION:
The purpose of this study is to assess and compare the overall efficacy and differential effects of two interventions for patients suffering from obsessive-compulsive disorder (OCD) according to DSM-5. The interventions to be compared are detached mindfulness (DM) and cognitive restructuring (CR). Whereas the efficacy of CR for the treatment of OCD has been proven in various studies, the efficacy of DM as a single intervention so far has only been shown within a case study and within a non-clinical sample. By contrast, the efficacy of complex metacognitive protocols (of which DM constitutes one of several single interventions) has been shown multiple times. So far, however, little is known about the efficacy of DM as a single intervention in a clinical sample and the differential working mechanisms of DM vs. CR.

Whereas DM is supposed to modify metacognitions by teaching patients to solely observe their intrusive thoughts, CR aims at teaching the patients to actively question and modify their distorted interpretations of their intrusions. Since previous research has shown that symptom reduction is mediated by a change in metacognition but not by a change of distorted interpretations, the investigators hypothesize that, while expecting both interventions to be similarly effective on an overall scale, DM will lead to a change in both metacognitions and distorted interpretations whereas CR will predominantly have an effect on distorted interpretations while influencing metacognitions to a lesser extent. Further research questions address differences concerning the applicability of the two interventions in patients' everyday life and the degree to which an intense psychoeducation can already have an effect on the participants' overall symptom burden.

The intervention (both DM and CR) is spread over four sessions of 100 min each taking place within two weeks (i.e. two sessions per week) and includes intensive homework assignments for the patients. The intervention will be delivered by MSc-level clinical psychologists completing the clinical training for becoming a licenced psychotherapist in Germany ("Psychologischer Psychotherapeut"). The diagnostic assessment involves clinical interviews and a number of questionnaires and will be conducted by independent assessors who have a qualification similar to the study therapists. Assessment involves pre-, post- and follow-up assessment. Additionally, assessment comprises data collection via ecological momentary assessment (EMA) in order to measure OCD symptoms (intrusions, emotions and coping strategies), the degree to which participants apply the newly learned strategy (DM or CR) in everyday life and the amount of relief experienced from applying it. There will be one EMA before (Pre-EMA) and one after the intervention (Post-EMA). For EMA, participants receive a smartphone for four days each (Friday to Monday) and are randomly prompted ten times per day to fill in a short questionnaire. The average amount of time necessary to fill in the questionnaire is assumed to be less than 2 min, based on a sample trial with mentally healthy participants.

Participants will be randomly assigned to one of three groups: 1) DM, 2) CR, and 3) a waitlist control group. The waitlist control group will wait for two weeks (i.e., as long as the intervention in the other two groups last), before participants will be once more randomly assigned to one of the two active conditions (DM and CR), which they will then regularly participate in. Thus, all participants enrolled in the study receive one of the two treatments sooner or later. For participants who are initially assigned to the waitlist group, there will be a second pre-assessment prior to the start of the intervention.

The study is going to be sponsored by the Christoph-Dornier-Stiftung für Klinische Psychologie, which is a non-profit organization that supports research in clinical psychology and awards PhD scholarships to clinical psychologists. The study at hand is the major part of the PhD project of Christian Rupp, M. Sc., and Charlotte Juergens, M. Sc., who are currently holding a PhD scholarship by the Christoph-Dornier-Stiftung für Klinische Psychologie. The Christoph-Dornier-Stiftung für Klinische Psychologie collaborates with Department of Clinical Psychology at the University of Muenster (Westfälische Wilhelms-Universität). The The PhD project is being supervised scientifically by Principal Investigator Prof. Dr. Ulrike Buhlmann, who is a professor of clinical psychology at the University of Muenster (Westfälische Wilhelms-Universität), Germany.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of OCD according to DSM-5
* Minimum age of 18 years
* Sufficient German language skills

Exclusion Criteria:

* A mental disorder other then OCD constituting the primary diagnosis (such as depression)
* Verbal IQ <80 as measured with the MWT-B (Lehrl, 2005)
* Presence of an acute suicidal tendency or suicidal behavior in the past 6 months
* Presence of an acute psychosis or assured diagnosis of psychosis and related disorders
* Presence of an acute manic episode
* Presence of an acute borderline personality disorder
* Presence of a comorbid addictive disorder
* Present psychotherapeutic treatment including OCD-focused CBT elements
* Psychotherapeutic treatment including OCD-focused CBT elements within the past 12 months
* For individuals with psychotropic medication, a change of substance or dose within the past 8 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2018-07-12 (Actual); Study Completion 2018-07-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ulrike Buhlmann, Prof. Dr., Principal Investigator — Universität Münster
Locations (1):
- Christoph-Dornier-Stiftung für Klinische Psychologie, Münster, North Rhine-Westphalia, Germany

REFERENCES:
- [Background] Myers SG, Fisher PL, Wells A. An empirical test of the metacognitive model of obsessive-compulsive symptoms: fusion beliefs, beliefs about rituals, and stop signals. J Anxiety Disord. 2009 May;23(4):436-42. doi: 10.1016/j.janxdis.2008.08.007. Epub 2008 Sep 3. PMID 18922674
- [Background] Solem S, Haland AT, Vogel PA, Hansen B, Wells A. Change in metacognitions predicts outcome in obsessive-compulsive disorder patients undergoing treatment with exposure and response prevention. Behav Res Ther. 2009 Apr;47(4):301-7. doi: 10.1016/j.brat.2009.01.003. Epub 2009 Jan 17. PMID 19203749
- [Background] Gonner S, Leonhart R, Ecker W. [The German version of the obsessive-compulsive inventory-revised: a brief self-report measure for the multidimensional assessment of obsessive-compulsive symptoms]. Psychother Psychosom Med Psychol. 2007 Sep-Oct;57(9-10):395-404. doi: 10.1055/s-2007-970894. German. PMID 17590836
- [Background] Baer L. Alles unter Kontrolle: Zwangsgedanken und Zwangshandlungen überwinden. Bern: Hans Huber, 1993.
- [Background] Ertle A, Wahl K, Bohne A, Moritz S, Kordon A, Schulte D. Dimensionen zwangsspezifischer Einstellungen: Der Obsessive-Beliefs Questionnaire (OBQ) für den deutschen Sprachraum analysiert. Zeitschrift für Klinische Psychologie und Psychotherapie 37: 263-271, 2008.
- [Background] Hand I, Büttner-Westphal H. Die Yale-Brown Obsessive Compulsive Scale (Y-BOCS): Ein halbstrukturiertes Interview zur Beurteilung des Schweregrades von Denk- und Handlungszwängen. Verhaltenstherapie 1: 223-225, 1991.
- [Background] Wells A, Gwilliam P, Cartwright-Hatton S. Thought-Fusion-Instrument (TFI, unpublished manuscript). University of Manchester, UK, 2002.
- [Background] Schulte D. Messung der Therapieerwartung und Therapieevaluation von Patienten (PATHEV). Zeitschrift für Klinische Psychologie und Psychotherapie 34(3): 176-187, 2005.
- [Background] Hautzinger M, Keller F, Kühner C. BDI II. Beck Depressions Inventar. Revision. Frankfurt/Main: Harcourt Test Service, 2006.
- [Background] Wells A, McNicol K. Beliefs About Rituals Inventory (BARI, unpublished manuscript). University of Manchester, UK, 2004.
- [Background] Wells A. Metacognitive therapy for anxiety and depression. Guilford press, 2011.
- [Background] Wilhelm S, Steketee GS. Cognitive therapy for obsessive compulsive disorder: A guide for professionals. New Harbinger Publications, 2006.
- [Background] American Psychiatric Association. Diagnostic and statistical manual of mental disorders, Fourth Edition, Text Revision (DSM-IV-TR). Washington, DC: American Psychiatric Association, 2000.
- [Background] Wittchen HU, Wunderlich U, Gruschwitz S, Zaudig M. SKID I. Strukturiertes Klinisches Interview für DSM-IV. Achse I: Psychische Störungen. Interviewheft und Beurteilungsheft. Eine deutschsprachige, erweiterte Bearb. d. amerikanischen Originalversion des SKID I., 1997.
- [Background] Lehrl S. MWT-B Mehrfachwahl-Wortschatz-Intelligenztest. Balingen: Spitta-Verlag, 2005.
- [Background] Rosa-Alcazar AI, Sanchez-Meca J, Gomez-Conesa A, Marin-Martinez F. Psychological treatment of obsessive-compulsive disorder: a meta-analysis. Clin Psychol Rev. 2008 Dec;28(8):1310-25. doi: 10.1016/j.cpr.2008.07.001. Epub 2008 Jul 4. PMID 18701199
- [Background] Wilhelm S, Steketee G, Fama JM, Buhlmann U, Teachman BA, Golan E. Modular Cognitive Therapy for Obsessive-Compulsive Disorder: A Wait-List Controlled Trial. J Cogn Psychother. 2009;23(4):294-305. doi: 10.1891/0889-8391.23.4.294. PMID 21072138
- [Background] Olatunji BO, Rosenfield D, Tart CD, Cottraux J, Powers MB, Smits JA. Behavioral versus cognitive treatment of obsessive-compulsive disorder: an examination of outcome and mediators of change. J Consult Clin Psychol. 2013 Jun;81(3):415-28. doi: 10.1037/a0031865. Epub 2013 Feb 18. PMID 23421734
- [Background] Belloch A, Cabedo E, Carrio C, Larsson C. Cognitive therapy for autogenous and reactive obsessions: clinical and cognitive outcomes at post-treatment and 1-year follow-up. J Anxiety Disord. 2010 Aug;24(6):573-80. doi: 10.1016/j.janxdis.2010.03.017. Epub 2010 Apr 2. PMID 20418053
- [Background] Fisher PL, Wells A. Metacognitive therapy for obsessive-compulsive disorder: a case series. J Behav Ther Exp Psychiatry. 2008 Jun;39(2):117-32. doi: 10.1016/j.jbtep.2006.12.001. Epub 2007 Mar 7. PMID 17418090
- [Background] Rees CS, van Koesveld KE. An open trial of group metacognitive therapy for obsessive-compulsive disorder. J Behav Ther Exp Psychiatry. 2008 Dec;39(4):451-8. doi: 10.1016/j.jbtep.2007.11.004. Epub 2008 Jan 18. PMID 18295186
- [Background] Simons M, Schneider S, Herpertz-Dahlmann B. Metacognitive therapy versus exposure and response prevention for pediatric obsessive-compulsive disorder. A case series with randomized allocation. Psychother Psychosom. 2006;75(4):257-64. doi: 10.1159/000092897. PMID 16785776
- [Background] Shareh H, Gharraee B, Atef-Vahid MK, Eftekhar M. Metacognitive therapy (MCT), fluvoxamine, and combined treatment in improving obsessive-compulsive, depressive and anxiety symptoms in patients with obsessive-compulsive disorder (OCD). Iranian Journal of Psychiatry and Behavioral Sciences, 4(2): 17-25, 2010.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited between December 2016 and June 2018.
Groups:
- Detached Mindfulness: Group of patients receiving detached mindfulness (for details, see detailed description of the study)
- Cognitive Restructuring: Group of patients receiving cognitive restructuring (for details, see detailed description of the study)
- Waitlist: Group of patients who are re-randomized to either Detached Mindfulness or Cognitive Restructuring after a delay of 2 weeks.
Period: First Randomization
Arm/Group | Detached Mindfulness | Cognitive Restructuring | Waitlist
Started | 10 | 12 | 21
Completed | 9 | 11 | 21
Not Completed | 1 | 1 | 0
Period: Second Randomization (Re-randomization)
Arm/Group | Detached Mindfulness | Cognitive Restructuring | Waitlist
Started | 11 | 10 | 0
Completed | 11 | 9 | 0
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Please note that in contrast to the previous version of this document, we now listed the data for the intention-to-treat (ITT) sample, which is n = 43 (DM: n = 21, CR: n = 22), whereas the completer sample is n = 40 (DM: n = 20, CR: n = 20). We chose to do this because we also report the ITT sample in the article submitted for publication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Detached Mindfulness | Cognitive Restructuring | Total
Number analyzed (Participants) | 21 | 22 | 43
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.81 (9.48) | 31.23 (10.96) | 31.02 (10.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 10 | 25
  Male | 6 | 12 | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 21 | 22 | 43
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 21 | 22 | 43
Number of participants under parallel psychopharmacological medication [Count of Participants; unit: Participants] | 8 | 11 | 19

OUTCOME MEASURES:

1. Primary Outcome: Y-BOCS Change Score (Pre to Post Assessment)
Description: German version of the Yale-Brown Obsessive Compulsive Scale (Hand & Büttner-Westphal, 1991). The mininum value is 0, the maximal value is 40. Higher scores indicate a higher symptom severity of obsessive-compulsive disorder.
Time Frame: Difference score resulting from (a) first baseline minus post-treatment (non-waitlist) or (b) first baseline minus second baseline (waitlist). In both cases, there are 2 weeks between the two measurements.
Population: People with obsessive-compulsive disorder
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Waitlist: Waitlist control group, which, however, is again randomized after the waiting time in order to receive one of the two interventions (DM or CR).
Arm/Group | Detached Mindfulness | Cognitive Restructuring | Waitlist
Number analyzed (Participants) | 9 | 11 | 20
units on a scale | 5.11 (5.80) | 5.09 (5.43) | 0.25 (2.15)

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed because this trial eomployed a purely behavioral intervention for obsessive-compulsive disorder which from our point of view did not imply any potential side effects leading to a participant's death.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed because this trial eomployed a purely behavioral intervention for obsessive-compulsive disorder which from our point of view did not imply any potential side effects leading to a participant's death.
Groups:
- Detached Mindfulness (DM): Group of patients receiving detached mindfulness (for details, see detailed description of the study)
- Cognitive Restructuring (CR): Group of patients receiving cognitive restructuring (for details, see detailed description of the study)
- Waitlist (WL): Waitlist control group, which, however, is again randomized after the waiting time in order to receive one of the two interventions (DM or CR).
Arm/Group | Detached Mindfulness (DM) | Cognitive Restructuring (CR) | Waitlist (WL)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2018-07-12): https://cdn.clinicaltrials.gov/large-docs/53/NCT03002753/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-12): https://cdn.clinicaltrials.gov/large-docs/53/NCT03002753/SAP_001.pdf